CLINICAL TRIAL: NCT07027475
Title: Prospective Clinical Registry of Acute Treatment and Long-term Assessment of Adults Meningitis
Brief Title: Acute Treatment and Long-term Assessment of Adult Infectious Meningitis
Acronym: ATLAS-I
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: ATLAS-I
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Viral Meningitis; Bacterial Meningitis; Fungal Meningitis; Meningitis
Keywords: Meningitis; Bacterial; Viral; Corticosteroids; Antibiotics; Fungal
MeSH Terms: conditions — Meningitis, Viral; Meningitis, Bacterial; Meningitis, Fungal; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — cerebrospinal fluid, blood (serum)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multicenter, observational clinical registry of adult patients with acute infectious meningitis across approximately 30 public and private hospitals in Brazil. The study will include adults, 18 years old and older, with suspected acute infectious meningitis. Data will be collected during hospitalization and post-discharge to evaluate clinical management, treatment and short and long-term outcomes. The study aims to generate real-world evidence on current practices and outcomes to support improvements in national care protocols.

DETAILED DESCRIPTION:
This is a middle-income real-world prospective clinical registry study. Clinical and laboratory data will be collected during hospitalization and follow-up visits after discharge.

Data collection will include empirical antibiotic therapy timing and type, time from hospital admission to antibiotic's first dose, corticosteroid therapy initiation, vaccination status per the Brazilian National Immunization Program, neurological sequelae and access to specialized rehabilitation services post-discharge.

Primary outcomes will be all-cause mortality, length of hospital stay, rate of re- hospitalization and sensorineural hearing loss incidence.

Secondary outcomes will be etiology-specific mortality, functional outcomes (measured by modified Rankin Score and Barthel Index Brazilian version), guideline-based therapies by etiology, neurological sequelae incidence stratified by etiology (e.g., motor deficits, cerebrovascular complications) , serious adverse events and access to rehabilitation.

Findings will be used to inform public health system and clinical care in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Fever (axillary temperature ≥37.8°C) followed by two or more of the following symptoms: severe headache, vomiting, altered consciousness (confusion, drowsiness, or irritability), photophobia (increased sensitivity to light), presence of seizures OR
* Fever accompanied by at least one meningeal irritation sign, such as neck stiffness, Kernig's sign, or Brudzinski's sign OR
* Sudden onset of fever and appearance of petechial skin rash or hemorrhagic suffusions

Exclusion Criteria:

- Refusal to provide consent for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, ≥ 18 years old, suspect acute meningitis infection
Sampling Method: Probability Sample
Enrollment: 624 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mortality, re-hospitalization, length of hospital stay and sensory hearing loss | Day 28
  The primary outcome is a composite endpoint that includes:
  Incidence of all-cause death Incidence of all-cause re-hospitalization Length of initial hospital stay (measured in days) Incidence of sensory hearing loss

SECONDARY OUTCOMES:
Patients with guideline-directed therapy | Day 180
  Proportion of patients receiving empirical and targeted therapies according to national meningitis management guidelines
Mortality in six months | Day 180
  Incidence of all-cause mortality
Length of hospitalization by etiology | Day 180
  Length of hospitalization (in days), stratified by infectious etiology
Re-hospitalization rate | Day 180
  Rate of all-cause re-hospitalization
Invasive ventilatory support | Day 28
  Incidence of invasive ventilatory support
Access to specialized rehabilitation services | Day 180
  Proportion of patients receiving specialized rehabilitation care
Re-hospitalization rate by etiology | Day 180
  Rate of unplanned re-hospitalization stratified by etiology
Neurological sequelae by etiology | Day 180
  Incidence of neurological sequelae stratified by etiology
Post-discharge functional decline | Day 180
  Functional status decline assessed on follow-up using Functional independence measured by modified Rankin Score ≤ 2 and Barthel Index (Brazilian version)
  Functional status will be assessed using two standardized measures: the Modified Rankin Score (mRS) and the Barthel Index (Brazilian version). Decline in functional independence will be categorized as follows:
  * Mild disability: defined by an mRS score of 0 to 2 and a Barthel Index score of 90 or higher, indicating independence or slight dependence in daily activities.
  * Moderate disability: defined by an mRS score of 3 and a Barthel Index score between 60 and 89, corresponding to moderate dependence requiring some assistance.
  * Severe disability: defined by an mRS score of 4-5 and a Barthel Index score below 60, reflecting severe dependence or bedridden status with the need for constant care.
Adverse Events | Day 28
  Incidence of adverse events
Adverse outcomes requiring secondary intervention by etiology | Day 180
  Incidence of adverse outcomes by etiology

CONTACTS AND LOCATIONS:
Overall Officials: Henrique A Fonseca, MD, PhD, Study Chair — Hospital Israelita Albert Einstein; Anna M Gomes, MD, Principal Investigator — Hospital Israelita Albert Einstein

IPD SHARING:
Plan to Share IPD: No